CLINICAL TRIAL: NCT05365490
Title: Post-approval Study of Transcarotid Artery Revascularization in Standard Risk Patients With Significant Carotid Artery Disease. The ROADSTER 3 Study
Brief Title: Post-approval Study of Transcarotid Artery Revascularization in Standard Risk Patients With Significant Carotid Artery Disease
Status: Completed | Type: Observational
Sponsor: Silk Road Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: SRM-2022-01
Record Dates: First submitted 2022-05-03; First posted 2022-05-09 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Carotid Artery Diseases
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Standard-risk patients requiring carotid intervention: Symptomatic or asymptomatic patients with a discrete lesion located in the internal carotid artery (ICA) with or without involvement of the contiguous common carotid artery (CCA), who require carotid artery revascularization.
  Interventions: Procedure: Transcarotid Artery Revascularization (TCAR)

INTERVENTIONS:
Procedure: Transcarotid Artery Revascularization (TCAR) — Carotid artery revascularization treated with the FDA-cleared ENROUTE Transcarotid NPS in conjunction with the FDA-approved ENROUTE Transcarotid Stent
  Other Names: Carotid Revascularization; Carotid Artery Stenting

SUMMARY:
The study objective is to evaluate real world usage of the ENROUTE Transcarotid Stent when used with the ENROUTE Transcarotid Neuroprotection System in patients at standard risk for adverse events from carotid endarterectomy

DETAILED DESCRIPTION:
This is an open label, single arm, multi-center post-approval study for the treatment of patients at standard risk for adverse events from carotid endarterectomy who require carotid revascularization and who are eligible for treatment using the ENROUTE Transcarotid Stent System and the ENROUTE Transcarotid Neuroprotection System. The study will enroll a maximum of 400 patients treated per protocol at 30-60 sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a discrete lesion located in the internal carotid artery (ICA) with or without involvement of the contiguous common carotid artery (CCA) determined by duplex ultrasound, CT/CTA, MR/MRA or angiography.
2. Patient must meet one of the following criteria regarding neurological symptom status and degree of stenosis:

   Symptomatic: ≥70% stenosis of the common or internal carotid artery by ultrasound or ≥50% stenosis of the common or internal carotid artery by angiogram

   OR

   Asymptomatic: ≥70% stenosis of the common or internal carotid artery by ultrasound or ≥60% stenosis of the common or internal carotid artery by angiogram
3. Target vessel must meet all requirements for ENROUTE Transcarotid Neuroprotection System and ENROUTE Stent System (refer to IFU for requirements).
4. Patient is ≥18 and <80 years of age.
5. Patient understands the nature of the procedure and has provided a signed informed consent using a form that has been reviewed and approved by the Institutional Review Board of the respective clinical site prior to the study procedure. This will be obtained prior to participation in the study.
6. Patient is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations.

Exclusion Criteria:

1. Patient meets any of the surgical high-risk criteria listed below.

   1. Anatomic high risk exclusion criteria:

      * Contralateral carotid artery occlusion
      * Tandem stenoses in the ICA >70% diameter reducing
      * High cervical carotid artery stenosis above the C2 vertebra
      * Restenosis after prior ipsilateral carotid endarterectomy
      * Bilateral carotid artery stenosis requiring treatment within 30 days after index procedure
      * Hostile Necks including prior neck irradiation, radical neck dissection, and cervical spine immobility
   2. Clinical high risk exclusion criteria:

      * Patient is ≥80 years of age
      * Patient has ≥2-vessel coronary artery disease (or has had revascularization procedure within the last 30 days) and/or angina
      * Patient has history of unresolved angina - Canadian Cardiovascular Society (CCS) angina class 3 or 4 OR unstable angina
      * Patient has congestive heart failure (CHF) - New York Heart Association (NYHA) Functional Class III or IV
      * Patient has a known severe left ventricular dysfunction - LVEF <30%
      * Patient has had a myocardial infarction within 6 weeks prior to the procedure
      * Patient has severe obstructive pulmonary disease (COPD) with either:

        * FEVI <50% predicted OR
        * chronic oxygen therapy OR
        * resting PO2 of ≤60 mmHG (room air)
      * Patient has permanent contralateral cranial and/or laryngeal nerve injury
      * Patient has chronic renal insufficiency (serum creatinine ≥2.5 mg/dL) or is on dialysis
2. Patient has an alternative source of cerebral embolus, including but not limited to:

   1. Chronic atrial fibrillation.
   2. Any episode of paroxysmal atrial fibrillation within the past 6 months, or history of paroxysmal atrial fibrillation requiring chronic anticoagulation.
   3. Knowledge of cardiac sources of thrombus. (If patient has left ventricular aneurysm, intracardiac filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcific aortic stenosis, endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma AND there is no confirmed thrombus on an echocardiogram performed within 3 months prior to index procedure, the patient may be eligible for enrollment).
   4. Recently implanted heart valve (either surgically or endovascularly) within 60 days prior to index procedure with confirmed emboli on echocardiogram.
   5. Abnormal angiographic findings: ipsilateral intracranial or extracranial arterial stenosis (as determined by pre-procedure angiography or CTA/MRA ≤6 months prior to index procedure) greater in severity than the lesion to be treated, cerebral aneurysm >5 mm, AVM (arteriovenous malformation) of the cerebral vasculature, or other abnormal angiographic findings.
3. Patient has a history of spontaneous intracranial hemorrhage within the past 12 months or has had a recent (<7 days) stroke of sufficient size (on CT or MRI) to place him or her at risk of hemorrhagic conversion during the procedure.
4. Patient had hemorrhagic transformation of an ischemic stroke within the past 60 days.
5. Patient with a history of major stroke prior to the TCAR procedure attributable to either carotid artery (CVA or retinal embolus) with major neurological deficit (NIHSS ≥5 OR mRS ≥3) likely to confound study endpoints 1 month after the TCAR procedure (because the deficit persists post-operatively).
6. Patient has an intracranial tumor.
7. Patient has an evolving stroke.
8. Patient has neurologic illnesses within the past 2 years characterized by fleeting or fixed neurologic deficit which cannot be distinguished from TIA or stroke, including but not limited to: moderate to severe dementia, partial or secondarily generalized seizures, complicated or classic migraine, tumor or other space-occupying brain lesions, subdural hematoma, cerebral contusion or other post-traumatic lesions, intracranial infection, demyelinating disease, or intracranial hemorrhage.
9. Patient has had a TIA or amaurosis fugax within 48 hrs. prior to the procedure
10. Patient has an isolated hemisphere
11. Patient had or will have open heart (e.g., CABG), endovascular stent procedure, valve intervention, vascular surgery, other major operation within 30 days of the index procedure.
12. Presence of a previous placed intravascular stent in target vessel or ipsilateral CCA or significant CCA inflow lesion.
13. Occlusion or [Thrombolysis in Myocardial Infarction Trial (TIMI 0)] "string sign" >1cm of the ipsilateral common or internal carotid artery.
14. An intraluminal filling defect (defined as an endoluminal lucency surrounded by contrast, seen in multiple angiographic projections, in the absence of angiographic evidence of calcification) whether or not it is associated with an ulcerated target lesion.
15. Ostium of CCA requires revascularization.
16. Patient has an open stoma in the neck.
17. Female patients who are pregnant or may become pregnant.
18. Patient has history of intolerance or allergic reaction to any of the study medications or stent materials (refer to ENROUTE stent IFU), including aspirin (ASA), ticlopidine, clopidogrel, statin or contrast media (that cannot be pre-medicated). Patients must be able to tolerate statins (or a permitted non-statin substitute) and a combination of ASA and ticlopidine or ASA and clopidogrel or alternative P2Y12 inhibitor..
19. Patient has a life expectancy <5 years without contingencies related to other medical, surgical, or interventional procedures or is at High Risk as per the Wallaert Score. Estimation of life expectancy and scoring per the Wallaert Score is to be performed prior to enrollment.
20. Patient has primary, recurrent or metastatic malignancy and does not have independent assessment of life expectancy of ≥5 years performed by the treating oncologist or an appropriate specialist other than the physician performing TCAR.
21. Patient has an unresolved/uncorrected bleeding disorder.
22. Patient has a known allergy to nitinol
23. Patient is known to have an active SARS-CoV-2 infection (Coronavirus-19 [COVID-19]) or has been previously diagnosed with COVID-19 with neurological sequelae that could confound endpoint assessments (e.g., baseline mRS>3).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with discrete lesion located in the internal carotid artery (ICA) with or without involvement of the contiguous common carotid artery (CCA) determined by duplex ultrasound, CT/CTA, MR/MRA or angiography.
  -Symptomatic: ≥70% stenosis of the common or internal carotid artery by ultrasound or ≥50% stenosis of the common or internal carotid artery by angiogram
  Or
  -Asymptomatic: ≥70% stenosis of the common or internal carotid artery by ultrasound or ≥60% stenosis of the common or internal carotid artery by angiogram
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Hierarchical composite of Major Adverse Events (MAEs) | within 30 days of the index procedure
  Hierarchical composite of Major Adverse Events (MAEs) defined as any death, stroke, or myocardial infarction within 30 days of the index procedure
Ipsilateral Stroke | within 31 to 365 days following the index procedure
  Ipsilateral stroke within 31 days to 365 days following the index procedure

SECONDARY OUTCOMES:
Incidence of cranial nerve injury | within 30 days of the index procedure
  Incidence of cranial nerve injury within 30 days of the index procedure
Stroke | within 30 days of the index procedure
  Stroke within 30 days of the index procedure
Death | within 30 days of the index procedure
  Death within 30 days of the index procedure
MI | within 30 days of the index procedure
  MI within 30 days of the index procedure
Stroke/Death/MI | within 30 days of the index procedure
  Stroke/Death/MI within 30 days of the index procedure
Ipsilateral Stroke | 31-365 days
  Ipsilateral stroke within 31 to 365 days of the index procedure
Persistent cranial nerve injury | at 6 months and 1 year
  Persistent cranial nerve injury at 6 months and 1 year
Rate of hierarchical ipsilateral stroke, death, and myocardial infarction | within 30 days of the index procedure
  Rate of hierarchical ipsilateral stroke, death, and myocardial infarction within 30 days of the index procedure
Cardiac death | 1 year
  Cardiac death at 1 year for patients who experienced an MI within 30 days of the index procedure
Access site complications | within 30 days of the index procedure
  Access site complications (arterial/venous)
Serious Hematoma/Bleeding complications | within 30 days of the index procedure
  Serious Hematoma/Bleeding complications (arterial/venous)
Rate of stent thrombosis or occlusion | within 30 days of the index procedure
  Rate of stent thrombosis or occlusion within 30 days of the index procedure
Rate of dissection | within 30 days of the index procedure
  Rate of dissection within 30 days of the index procedure (during index procedure or a reintervention procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Dermody, MD, Principal Investigator — Lancaster General Hospital; Jeffrey Jim, MD, Principal Investigator — Abbott Northwestern Minneapolis Heart Institute Foundation; Marc Schermerhorn, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (53):
- United States (53):
  - Valley Vascular Consultants, Huntsville, Alabama
  - HonorHealth, Scottsdale, Arizona
  - Pima Heart & Vascular, Tucson, Arizona
  - University of California, San Diego (UCSD), La Jolla, California
  - Sharp Grossmont, La Mesa, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Ocala, Ocala, Florida
  - Coastal Vascular & Interventional, Pensacola, Florida
  - Northside Vascular, Cumming, Georgia
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Carle Health, Urbana, Illinois
  - Deaconess Research / Evansville Surgical Associates, Evansville, Indiana
  - Indiana University, Indianapolis, Indiana
  - Baton Rouge General, Baton Rouge, Louisiana
  - Acadiana Vascular Clinic / Our Lady Lourdes Heart Hospital, Lafayette, Louisiana
  - Maine Medical Center, Portland, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - McLaren Heart & Vascular, Bay City, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Abbott Northwestern, Minneapolis, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Midwest Aortic & Vascular Institute, North Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York University, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke University, Raleigh, North Carolina
  - Bethesda North Hospital, Cincinnati, Ohio
  - St. Charles Health System, Bend, Oregon
  - Providence St. Vincent, Portland, Oregon
  - St. Luke's University Hospital, Bethlehem, Pennsylvania
  - UPMC Pinnacle, Harrisburg, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Stern Cardiovascular, Germantown, Tennessee
  - Cardiovascular Surgery Clinic, Memphis, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Baylor Scott & White Dallas, Dallas, Texas
  - Memorial Hermann Southeast, Houston, Texas
  - Baylor Scott & White Plano, Plano, Texas
  - Houston Methodist Sugarland, Sugarland, Texas
  - Sentara, Norfolk, Virginia
  - Carilion Roanoke Memorial, Roanoke, Virginia
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No
Not planning to share IPD

REFERENCES:
- [Background] Malas MB, Dakour-Aridi H, Kashyap VS, Eldrup-Jorgensen J, Wang GJ, Motaganahalli RL, Cronenwett JL, Schermerhorn ML. TransCarotid Revascularization With Dynamic Flow Reversal Versus Carotid Endarterectomy in the Vascular Quality Initiative Surveillance Project. Ann Surg. 2022 Aug 1;276(2):398-403. doi: 10.1097/SLA.0000000000004496. Epub 2020 Sep 15. PMID 32941280
- [Background] Schermerhorn ML, Liang P, Eldrup-Jorgensen J, Cronenwett JL, Nolan BW, Kashyap VS, Wang GJ, Motaganahalli RL, Malas MB. Association of Transcarotid Artery Revascularization vs Transfemoral Carotid Artery Stenting With Stroke or Death Among Patients With Carotid Artery Stenosis. JAMA. 2019 Dec 17;322(23):2313-2322. doi: 10.1001/jama.2019.18441. PMID 31846015
- [Background] Vilain KR, Magnuson EA, Li H, Clark WM, Begg RJ, Sam AD 2nd, Sternbergh WC 3rd, Weaver FA, Gray WA, Voeks JH, Brott TG, Cohen DJ; CREST Investigators. Costs and cost-effectiveness of carotid stenting versus endarterectomy for patients at standard surgical risk: results from the Carotid Revascularization Endarterectomy Versus Stenting Trial (CREST). Stroke. 2012 Sep;43(9):2408-16. doi: 10.1161/STROKEAHA.112.661355. Epub 2012 Jul 19. PMID 22821614